CLINICAL TRIAL: NCT02656017
Title: Metformin as a Novel Therapy for Autosomal Dominant Polycystic Kidney Disease
Acronym: TAME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyongtae Ty Bae, M.D., Ph.D. (Other)
Collaborators: Tufts Medical Center (Other); University of Maryland, Baltimore (Other); University of Southern California (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Kyongtae Ty Bae, M.D., Ph.D., Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO15060422; CDMRP-PR141606 (Other: US Army Medical Research and Materiel Command)
Record Dates: First submitted 2015-12-23; First posted 2016-01-14 (Estimated); Results first posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Polycystic Kidney, Autosomal Dominant
Keywords: kidney disease; polycystic kidney disease; autosomal dominant kidney disease; kidney cysts; PKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Kidney Diseases; Polycystic Kidney Diseases | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Participants will be started on 500 mg of metformin once daily, with the following scheduled dose titrations:
  * Increase to 500mg twice daily at week 2
  * Increase to 1000mg qAM, 500mg qPM at week 4
  * Increase to 1000mg twice daily at week 6 for the duration of their participation (26 months).
    * Increased titrations based on tolerability
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Participants will be started on 500 mg of placebo once daily, with the following scheduled dose titrations:
  * Increase to 500mg twice daily at week 2
  * Increase to 1000mg qAM, 500mg qPM at week 4
  * Increase to 1000mg twice daily at week 6 for the duration of their participation (26 months).
    * Increased titrations based on tolerability
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metformin — Monitoring of tolerability and symptoms.
  Other Names: Glucophage; Metformin hydrochloride
  Arms: Metformin
Other: Placebo — Monitoring of tolerability and symptoms.
  Arms: Placebo

SUMMARY:
This study will test to see if metformin is safe and if it is tolerated compared to placebo in adult Autosomal Dominant Polycystic Kidney Disease (ADPKD) patients with beginning stages of chronic kidney disease. We will also measure its effect on progression of kidney disease as reflected in the kidney size and the kidney function, along with its effect on kidney pain and quality of life.

DETAILED DESCRIPTION:
There is growing evidence that metformin, a drug widely used for the treatment of type 2 diabetes and polycystic ovary syndrome, may serve as a novel therapy for individuals in the early stages of Autosomal Dominant Polycystic Kidney Disease ADPKD by activating the metabolic sensor AMP-activated protein kinase (AMPK). AMPK is activated under conditions of metabolic and other cellular stresses. Through its actions on downstream mediators, AMPK activation during low energy states decreases cellular energy consumption while stimulating energy generating pathways. It has been shown that AMPK phosphorylates and inhibits cystic fibrosis transmembrane conductance regulator (CFTR), thus suppressing epithelial fluid and electrolyte secretion. Similarly, AMPK phosphorylates the tuberin protein, leading to indirect inhibition of the mTOR pathway. Thus, AMPK inhibits both CFTR and mTOR, suggesting that targeted activation of this kinase by metformin may provide a therapeutic benefit in ADPKD. It has been shown that metformin treatment of kidney epithelial cells leads to stimulation of AMPK and subsequent inhibition of both mTOR and CFTR activity. It has also been shown that metformin slows cystogenesis in animal models of PKD, supporting the potential of this drug in ADPKD treatment.

ELIGIBILITY:
Inclusion Criteria:

Subject has Autosomal Dominant Polycystic Kidney Disease; Subject is fluent in English

Exclusion Criteria:

Subject is not on active military duty; Subject is not currently participating in another clinical trial; Subject's current GFR is not <50 cc/min/1.73m2; Subject does not have diabetes; Subject does not have a systemic disease other than hypertension and PKD; Subject does not have a solitary kidney; Subject does not have an allergy or intolerance to metformin; Subject is not pregnant or lactating or intending to become pregnant within the next three years; Subject does not have an unstable or unclipped cerebral aneurysm; Subject does not have active coronary artery disease; Subject does not have an MRI incompatible device/implant; Subject does not have severe claustrophobia; Subject has not had any solid organ transplant; Subject does not have a Vitamin B12 deficiency; Subject does not currently take any medications that interact with metformin, such as nifedipine, furosemide, cationic drugs (amiloride, ranitidine, triamterene digoxin, procainamide, quinidine, vancomycin, trimethoprim); Subject does not currently take nor has taken (within 2 weeks) the drug tolvaptan (Jynarque or Samsca)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyongtae Bae, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Maryland Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] El-Damanawi R, Stanley IK, Staatz C, Pascoe EM, Craig JC, Johnson DW, Mallett AJ, Hawley CM, Milanzi E, Hiemstra TF, Viecelli AK. Metformin for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2024 Jun 4;6(6):CD013414. doi: 10.1002/14651858.CD013414.pub2. PMID 38837240
- [Derived] Seliger SL, Watnick T, Althouse AD, Perrone RD, Abebe KZ, Hallows KR, Miskulin DC, Bae KT. Baseline Characteristics and Patient-Reported Outcomes of ADPKD Patients in the Multicenter TAME-PKD Clinical Trial. Kidney360. 2020 Dec 31;1(12):1363-1372. doi: 10.34067/KID.0004002020. PMID 33768205

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Participants will be started on 500 mg of metformin once daily, with the following scheduled dose titrations:
  * Increase to 500mg twice daily at week 2
  * Increase to 1000mg qAM, 500mg qPM at week 4
  * Increase to 1000mg twice daily at week 6 for the duration of their participation (26 months).
    * Increased titrations based on tolerability
  Metformin: Monitoring of tolerability and symptoms.
- Placebo: Participants will be started on 500 mg of placebo once daily, with the following scheduled dose titrations:
  * Increase to 500mg twice daily at week 2
  * Increase to 1000mg qAM, 500mg qPM at week 4
  * Increase to 1000mg twice daily at week 6 for the duration of their participation (26 months).
    * Increased titrations based on tolerability
  Placebo: Monitoring of tolerability and symptoms.
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 49 | 48
Completed | 40 | 42
Not Completed | 9 | 6
Not completed — Study burden | 3 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Unable/unwilling to take study medication | 2 | 1
Not completed — Began Tolvaptan | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 48 | 97
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (10.4) | 42.1 (10.1) | 41.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 32 | 70
  Male | 11 | 16 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 8
  Not Hispanic or Latino | 47 | 42 | 89
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 46 | 46 | 92
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 49 | 48 | 97
PKD genotype [Count of Participants; unit: Participants]
  PKD1 | 37 | 28 | 65
  PKD2 | 7 | 10 | 17
  Other | 1 | 4 | 5
  No mutation detected | 2 | 4 | 6
  N/A | 2 | 2 | 4
GFR [Mean (Standard Deviation); unit: (ml/min/1.73 m²)] | 86.1 (20.6) | 85.9 (19.0) | 86.0 (19.7)
Vitamin B12 [Mean (Standard Deviation); unit: pg/mL] | 580.7 (350.8) | 495.3 (202.3) | 538.4 (288.8)
Glucose [Mean (Standard Deviation); unit: mg/dL] | 88.6 (8.4) | 90.9 (9.1) | 89.7 (8.8)
HbA1c [Mean (Standard Deviation); unit: % of total hemoglobin] — Population: Two participants are missing results.
  % of total hemoglobin
    number analyzed (Participants) | 48 | 47 | 95
    (all) | 5.2 (0.3) | 5.2 (0.3) | 5.2 (0.3)
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.92 (0.24) | 0.94 (0.23) | 0.93 (0.23)
Systolic BP [Mean (Standard Deviation); unit: mmHg] | 122.2 (13.1) | 124.1 (13.0) | 123.1 (13.0)
Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 76.8 (8.9) | 74.6 (8.5) | 75.7 (8.7)
Weight [Mean (Standard Deviation); unit: kg] | 78.5 (16.9) | 78.2 (17.4) | 78.4 (17.0)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.0 (5.9) | 26.6 (4.5) | 26.8 (5.2)
Gastrointestinal Symptoms Rating Scale [Mean (Standard Deviation); unit: scores on a scale] — GSRS is a widely used, validated 15-item questionnaire used to assess GI symptom burden (minimum, maximum: 1, 7, where higher mean score is worse outcome).
  scores on a scale | 1.4 (0.5) | 1.3 (0.4) | 1.4 (0.4)
Short Form-36, Mental Component Summary [Mean (Standard Deviation); unit: scores on a scale] — Short Form-36 Quality of Life Mental Component Summary (SF-36 MCS) ranges from 0 (worst possible outcome) to 100 (best possible outcome).
  scores on a scale | 51.7 (9.0) | 53.1 (7.9) | 52.4 (8.5)
Short Form-36, Physical Component Summary [Mean (Standard Deviation); unit: scores on a scale] — Short Form-36 Quality of Life Physical Component Summary (SF-36 PCS) ranges from 0 (worst possible outcome) to 100 (best possible outcome).
  scores on a scale | 52.2 (6.5) | 53.2 (6.3) | 52.7 (6.4)
Mayo Imaging Class [Count of Participants; unit: Participants] — For Measure Description: Imaging classification of ADPKD, where height-adjusted total kidney volume is stratified into classes on the basis of kidney size and age (class 2, 1A-1E, in increasing order of risk for eGFR decline).
  Participants
    Class 2 | 2 | 5 | 7
    Class 1A | 9 | 6 | 15
    Class 1B | 13 | 15 | 28
    Class 1C | 14 | 12 | 26
    Class 1D | 6 | 6 | 12
    Class 1E | 4 | 4 | 8
    N/A | 1 | 0 | 1
Height-adjusted total kidney volume [Mean (Standard Deviation); unit: mL/m] — Population: One participant missing result.
  mL/m
    number analyzed (Participants) | 48 | 48 | 96
    (all) | 625.8 (386.5) | 750.9 (547.8) | 688.4 (475.7)
Height-adjusted liver volume [Mean (Standard Deviation); unit: mL/m] — Population: One participant missing result.
  mL/m
    number analyzed (Participants) | 48 | 48 | 96
    (all) | 1,224.1 (490.7) | 1,019.0 (212.6) | 1,121.6 (390.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Gastrointestinal Symptoms Rating Scale (GSRS) to 24 Months
Description: GSRS is a widely used, validated 15-item questionnaire used to assess GI symptom burden (minimum, maximum: 1, 7, where higher mean score is worse outcome).
  Mean change to 24 months, estimated with a repeated measures analysis (baseline, 2 weeks, 6 weeks, 1 month, 3 months and every 3 months thereafter to 24 months) using a linear mixed model.
Time Frame: Baseline, 2 weeks, 6 weeks, 1 month, 3 months and every 3 months thereafter to 24 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 49 | 48
score on a scale | -0.04 [-0.18 to 0.10] | -0.11 [-0.24 to 0.03]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Linear mixed model with random intercept was used to compare the change in GSRS score as a function of time, the interaction between time and study arm, and clinical site; Test type: Superiority; p = 0.50, Mixed Models Analysis; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.13 to 0.26]

2. Primary Outcome: Drug Tolerability
Description: Tolerability was based on the first visit a participant responded no to the following question "Can you tolerate this dose of study drug the rest of your life?", which was asked at baseline, 2 weeks, 6 weeks, 1 month, 3 months and every 3 months thereafter to 24 months.
Time Frame: Baseline, 2 weeks, 6 weeks, 1 month, 3 months and every 3 months thereafter to 24 months
Population: Intention to treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 49 | 48
Participants | 21 | 14
Statistical Analysis 1: Comparison: Metformin vs Placebo; The Gray's test of homogeneity for competing risks was used to compare cumulative incidence of tolerating the drug between study arms; Test type: Superiority; p = 0.12, Gray's test

3. Primary Outcome: Rate of Serious Adverse Events (SAE)
Description: Serious adverse events (SAE) occurring from the time a participant signs the informed consent (at the screening visit) until the end of the study, meeting 1 or more of the criteria of: 1) Resulting in death, 2) Non-elective hospitalization, 3) Life threatening (if patient continued on study drug would result in death), 4) Harming or disabling persistently or permanently , 5) Exceeding the nature, severity or frequency of risk described in the protocol or 6) Resulting in congenital anomaly.
Time Frame: 26 months
Population: Participants who received and took metformin or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 49 | 48
Participants | 4 | 4
Statistical Analysis 1: Comparison: Metformin vs Placebo; Cumulative incidence between study arms and logistic regression was used to assess the association between study arms; Test type: Superiority; p = 0.98, Regression, Logistic

4. Secondary Outcome: Quality of Life Physical Component
Description: Short Form-36 Quality of Life Physical Component Summary (SF-36 PCS) ranges from 0 (worst possible outcome) to 100 (best possible outcome).
  Mean change to 24 months, estimated with a repeated measures analysis (baseline, 1 month, 3 months and every 3 months thereafter to 24 months) using a linear mixed model.
Time Frame: Baseline, 1 month, 3 months and every 3 months thereafter to 24 months
Population: Intention to treat analysis
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 49 | 48
score on a scale | -0.11 [-1.69 to 1.46] | -0.51 [-2.05 to 1.03]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Linear mixed model with random intercept was used to compare the change in SF-36 PCS as a function of time, the interaction between time and study arm, and clinical site; Test type: Superiority; p = 0.72, Mixed Models Analysis; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-1.81 to 2.60]

5. Secondary Outcome: Quality of Life Mental Component
Description: Short Form-36 Quality of Life Mental Component Summary (SF-36 MCS) ranges from 0 (worst possible outcome) to 100 (best possible outcome).
  Mean change to 24 months, estimated with a repeated measures analysis (baseline, 1 month, 3 months and every 3 months thereafter to 24 months) using a linear mixed model.
Time Frame: Baseline, 1 month, 3 months and every 3 months thereafter to 24 months
Population: Intention to treat analysis
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 49 | 48
score on a scale | 1.01 [-1.23 to 3.25] | -0.11 [-2.29 to 2.08]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Linear mixed model with random intercept was used to compare the change in SF-36 MCS as a function of time, the interaction between time and study arm, and clinical site; Test type: Superiority; p = 0.49, Mixed Models Analysis; Mean Difference (Final Values) = 1.11, 95% CI 2-sided [-2.02 to 4.25]

6. Secondary Outcome: Back Pain Frequency Over the Past 3 Months Since Last Visit
Description: Odds ratio (OR) per month of back pain Often, Usually, or Always (vs. Never, Rarely, Sometimes) estimated with a repeated measures analysis (baseline, 1 month, 3 months and every 3 months thereafter to 24 months) using a generalized linear mixed model.
Time Frame: Baseline, 1 month, 3 months and every 3 months thereafter to 24 months
Population: Intention to treat analysis
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 49 | 48
odds ratio | 0.95 [0.90 to 1.00] | 0.92 [0.88 to 0.98]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Generalized linear mixed model (logit link) with random intercept and slope was used to compare back pain frequency as a function of time, the interaction between time and study arm, and clinical site; Test type: Superiority; p = 0.44, Mixed Models Analysis

7. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: Mean change to 24 months, estimated with a repeated measures analysis (baseline, 2 weeks, 6 weeks, 1 month, 3 months and every 3 months thereafter to 24 months) using a linear mixed model.
Time Frame: Baseline, 2 weeks, and 6 weeks, 1 month, 3 months and every 3 months thereafter to 24 months
Population: Intention to treat analysis
Measure: Mean (95% Confidence Interval); unit: ml/min/1.73m^2
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 49 | 48
ml/min/1.73m^2 | -3.41 [-6.36 to -0.46] | -6.14 [-9.04 to -3.24]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Linear mixed model with random intercept was used to compare the change in eGFR as a function of time, the interaction between time and study arm, and clinical site; Test type: Superiority; p = 0.20, Mixed Models Analysis; Mean Difference (Final Values) = 2.73, 95% CI 2-sided [-1.40 to 6.87]

8. Secondary Outcome: Total Kidney Volume From Magnetic Resonance Imaging
Description: Annual percent change of height adjusted and natural log transformed total kidney volume [ln(htTKV)] was estimated with a linear mixed model.
Time Frame: Baseline, 6 months, 12 months, 18 months, 24 months
Population: Intention to treat analysis
Measure: Mean (95% Confidence Interval); unit: annual percent change
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 49 | 48
annual percent change | 3.87 [1.09 to 6.74] | 2.16 [-0.52 to 4.91]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Linear mixed model with random intercept and slope was used to compare the annual percent change of ln(htTKV) as a function of time, the interaction between time and study arm, and clinical site; Test type: Superiority; p = 0.38, Mixed Models Analysis; Mean Difference (Final Values) = 1.68, 95% CI 2-sided [-2.11 to 5.62]

9. Secondary Outcome: Total Kidney Cyst Volume From Magnetic Resonance Imaging
Description: Annual percent change of height adjusted and natural log transformed total kidney cyst volume [ln(htTKCV)] was estimated with a linear mixed model.
Time Frame: Baseline, 6 months, 12 months, 18 months, 24 months
Population: Intention to treat analysis
Measure: Mean (95% Confidence Interval); unit: annual percent change
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 49 | 48
annual percent change | 9.37 [3.82 to 15.22] | 5.36 [0.13 to 10.86]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Linear mixed model with random intercept and slope was used to compare the annual percent change of ln(htTKCV) as a function of time, the interaction between time and study arm, and clinical site; Test type: Superiority; p = 0.31, Mixed Models Analysis; Mean Difference (Final Values) = 3.81, 95% CI 2-sided [-3.48 to 11.65]

10. Secondary Outcome: Liver Volume From Magnetic Resonance Imaging
Description: Annual percent change of height adjusted and natural log transformed liver volume [ln(htLV)] was estimated with a linear mixed model.
Time Frame: Baseline, 6 months, 12 months, 18 months, 24 months
Population: Intention to treat analysis
Measure: Mean (95% Confidence Interval); unit: annual percent change
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 49 | 48
annual percent change | 1.60 [0.02 to 3.21] | 1.21 [-0.32 to 2.77]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Linear mixed model with random intercept and slope was used to compare the annual percent change of ln(htLV) as a function of time, the interaction between time and study arm, and clinical site; Test type: Superiority; p = 0.72, Mixed Models Analysis; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [-1.78 to 2.61]

11. Secondary Outcome: Liver Cyst Volume From Magnetic Resonance Imaging
Description: Annual percent change of height adjusted and natural log transformed liver cyst volume [ln(htLCV)] was estimated with a linear mixed model.
Time Frame: Baseline, 6 months, 12 months, 18 months, 24 months
Population: Intention to treat analysis
Measure: Mean (95% Confidence Interval); unit: annual percent change
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 49 | 48
annual percent change | 12.72 [3.47 to 22.79] | 10.94 [1.73 to 20.99]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Linear mixed model with random intercept and slope was used to compare the annual percent change of ln(htLCV) as a function of time, the interaction between time and study arm, and clinical site; Test type: Superiority; p = 0.80, Mixed Models Analysis; Mean Difference (Final Values) = 1.60, 95% CI 2-sided [-10.05 to 14.76]

12. Secondary Outcome: Frequency Abdominal Fullness Interfered With Ability to Perform Usual Physical Activity Over the Past 3 Months Since Last Visit.
Description: Odds ratio (OR) per month of abdominal fullness interfered Often, Usually, or Always (vs. Never, Rarely, Sometimes) estimated with a repeated measures analysis (baseline, 1 month, 3 months and every 3 months thereafter to 24 months) using a generalized linear mixed model.
Time Frame: Baseline, 1 month, 3 months and every 3 months thereafter to 24 months
Population: Intention to treat analysis
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 49 | 48
odds ratio | 1.00 [0.89 to 1.13] | 0.99 [0.87 to 1.12]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Generalized linear mixed model (logit link) with random intercept and slope was used to compare abdominal fullness interfered as a function of time, the interaction between time and study arm, and clinical site; Test type: Superiority; p = 0.83, Mixed Models Analysis

13. Secondary Outcome: Interference of Pain With Sleep Over the Past 3 Months Since Last Visit
Description: Odds ratio (OR) per month of pain interfered with sleep Quite a bit or Extremely (vs. Not at all, A little bit, Moderately) estimated with a repeated measures analysis (baseline, 1 month, 3 months and every 3 months thereafter to 24 months) using a generalized linear mixed model.
Time Frame: Baseline, 1 month, 3 months and every 3 months thereafter to 24 months
Population: Intention to treat analysis
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 49 | 48
odds ratio | 1.00 [0.87 to 1.14] | 0.97 [0.88 to 1.07]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Generalized linear mixed model (logit link) with random intercept and slope was used to compare interference of pain with sleep frequency as a function of time, the interaction between time and study arm, and clinical site; Test type: Superiority; p = 0.72, Mixed Models Analysis

14. Secondary Outcome: Interference of Pain With Strenuous Physical Activity Over the Past 3 Months Since Last Visit
Description: Odds ratio (OR) per month of pain interfered with strenuous physical activity Quite a bit or Extremely (vs. Not at all, A little bit, Moderately) estimated with a repeated measures analysis (baseline, 1 month, 3 months and every 3 months thereafter to 24 months) using a generalized linear mixed model.
Time Frame: Baseline, 1 month, 3 months and every 3 months thereafter to 24 months
Population: Intention to treat analysis
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 49 | 48
odds ratio | 0.99 [0.93 to 1.06] | 0.95 [0.90 to 1.01]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Generalized linear mixed model (logit link) with random intercept and slope was used to compare interference of pain with strenuous physical activity frequency as a function of time, the interaction between time and study arm, and clinical site; Test type: Superiority; p = 0.28, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse event were data collected at 2, 4, and 6 weeks during the titration period and every 3 months thereafter through 26 months.
Description: Adverse events and deaths were not collected by dose level.
Arm/Group | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/48
Serious Adverse Events (participants affected / at risk) | 4/49 | 4/48
Other Adverse Events (participants affected / at risk) | 21/49 | 13/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=49) | Placebo (N=48)
Other - diarrhea (c. difficile infection) (Infections and infestations) | 1 (1) | 0 (0)
Other - bone fracture (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Other - lightheadedness (Nervous system disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Other - umbilical hernia (Surgical and medical procedures) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Other - urinary tract infection and renal cyst hemorrhage (mild) (Infections and infestations) | 0 (0) | 1 (1)
Other - renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Other - renal cyst rupture (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=49) | Placebo (N=48)
Diarrhea (Gastrointestinal disorders) | 21 (42) | 13 (18)
Nausea (Gastrointestinal disorders) | 17 (29) | 10 (15)
Abdominal Pain (Gastrointestinal disorders) | 8 (11) | 9 (9)
Flatulence (Gastrointestinal disorders) | 10 (12) | 7 (7)
Constipation (Gastrointestinal disorders) | 6 (6) | 7 (7)
Abdominal Distension (Gastrointestinal disorders) | 7 (8) | 4 (4)
Vomiting (Gastrointestinal disorders) | 5 (6) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 3 (5) | 2 (2)
Bloating (Gastrointestinal disorders) | 5 (5) | 1 (1)
Other - Loss Of Appetite (Gastrointestinal disorders) | 2 (2) | 3 (4)
Other - Loose Stools (Gastrointestinal disorders) | 3 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 9 (11)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 7 (8)
Other - Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Hematuria (Renal and urinary disorders) | 3 (3) | 4 (4)
Other - Uti (Renal and urinary disorders) | 2 (3) | 3 (3)
Other - Kidney Pain (Renal and urinary disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 8 (11) | 6 (8)
Dizziness (Nervous system disorders) | 4 (4) | 3 (4)
Fatigue (General disorders) | 4 (4) | 5 (5)
Chills (General disorders) | 0 (0) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (5) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 4 (6) | 3 (4)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT02656017/Prot_SAP_001.pdf
  • Informed Consent Form (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT02656017/ICF_000.pdf